CLINICAL TRIAL: NCT01789567
Title: Engager Direct Aortic Clinical Study: Medtronic Engager™ Transcatheter Aortic Valve Implantation System Via Direct Aortic Approach
Brief Title: Engager Direct Aortic Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAE00807
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Results first posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2017-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Engager™ aortic valve (Other): Implantation of the Medtronic Engager™ bioprosthesis via direct aortic approach
  Interventions: Device: Engager™ aortic valve

INTERVENTIONS:
Device: Engager™ aortic valve — Implantation of the Medtronic Engager™ bioprosthesis via direct aortic approach

SUMMARY:
To confirm the safety and performance of the Medtronic Engager™ Transcatheter Aortic Valve Implantation System via direct aortic approach.

DETAILED DESCRIPTION:
To confirm the safety and performance of the Medtronic Engager™ Transcatheter Aortic Valve Implantation System via direct aortic approach in patients with symptomatic severe aortic valve stenosis at high or extreme risk for surgical aortic valve replacement for which treatment via direct aortic access is preferred.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis as defined by Doppler echocardiography: aortic valve area ≤ 0.8 cm2 (or AVA index ≤ 0.5 cm2/m2), or mean gradient ≥ 40 mmHg, or max velocity ≥ 4m/s
* NYHA Functional Class II or greater;
* Logistic EuroSCORE I ≥ 20%, or comorbidity judged by the heart team to pose an absolute or relative contraindication for conventional aortic valve replacement;
* Non-calcified ascending aortic site ≥ 50 mm from the aortic valve basal plane;
* Age ≥ 18 years;
* The patient has been informed of the nature of the study and has consented to participate, authorizing the collection and release of his/her medical information by signing a consent form ("Patient Informed Consent Form"). Patient should understand the implications of participating in the study and should be legally competent to provide informed consent.

Exclusion Criteria:

* Unicuspid or bicuspid aortic valve;
* Echocardiographic evidence of intracardiac mass, thrombus, or vegetation;
* Left ventricular ejection fraction < 25%;
* Left ventricular outflow obstruction, such as Hypertrophic Obstructive Cardiomyopathy and severe septal hypertrophy;
* Mitral or tricuspid regurgitation greater than 2+ by angiography or moderate by echocardiography;
* Patients with life expectancy less than 12 months due to an underlying non-cardiac co-morbid disease;
* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, Nitinol or contrast medium that cannot be adequately controlled with pre-medication;
* Sepsis or acute endocarditis;
* Blood dyscrasia such as acute anemia, leucopenia, or thrombocytopenia; bleeding diathesis, or coagulopathy;
* Renal insufficiency assessed by creatinine clearance < 20 ml/min and/or end-stage renal disease requiring chronic dialysis;
* Active peptic ulcer or GI bleeding within 3 months from the planned index procedure;
* Untreated clinically significant coronary artery disease requiring revascularization;
* Cardiogenic shock, suspected cardiogenic shock, or hemodynamic instability requiring inotropic support or mechanical heart assistance;
* Significant aortic disease, including abdominal and thoracic aortic aneurysm, defined as maximal luminal diameter of 5 cm or greater;
* Need for emergency surgery, cardiac or non-cardiac;
* History of myocardial infarction in the last 6 weeks;
* History of TIA or CVA in the last 6 months;
* Therapeutic invasive cardiac procedure, with the exception of BAV, performed within 30 days of the planned date of valve implantation, or 6 months in the case of drug-eluting stents;
* Pre-existing prosthetic heart valve or prosthetic ring in any position;
* Patent RIMA or pre-existing patent RIMA graft at direct aortic access site and/or trajectory;
* Patient refuses a blood transfusion;
* Pregnant or breastfeeding women;
* Patient is currently enrolled in another investigational device or drug trial that may influence the outcome of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Treede, MD, Principal Investigator — University Hospital Halle, Germany; David Holzhey, MD, Principal Investigator — Leipzig Heart Institute, Germany; Sabine Bleiziffer, MD, Principal Investigator — German Heart Center Munich, Germany; Marian Branny, MD, Principal Investigator — Nemocnice Podlesi, Trinec, Czech Republic; Neil Moat, MD, Principal Investigator — Royal Brompton Hospital, London, United Kingdom; Vinayak Bapat, MD, Principal Investigator — St. Thomas' Hospital, London, United Kingdom
Locations (6):
- Nemocnice Podlesí a.s., Třinec, Czechia
- Germany (3):
  - University Hospital Halle, Halle
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München, Munich
- United Kingdom (2):
  - St. Thomas' Hospital, London
  - Royal Brompton Hospital, London

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engager™ Aortic Valve
Started | 20
Completed | 14
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Engager™ Aortic Valve
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.6 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  Czech Republic | 3
  United Kingdom | 3
  Germany | 14
STS Risk of Mortality [Mean (Standard Deviation); unit: %] — The Society of Thoracic Surgeons (STS) Risk of Mortality model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables; scores are interpreted as follows: <4%, low risk; 4% to <8%, intermediate risk; 8% to <12%, high risk; ≥ 12%, very high risk.
  % | 5.9 (4.7)
Peripheral vascular disease [Number; unit: participants]
  Peripheral vascular disease | 10
  No peripheral vascular disease | 10

OUTCOME MEASURES:

1. Primary Outcome: Acute Delivery System Success
Description: Acute delivery system success, defined as bioprosthesis deployed in anatomically correct position and freedom from delivery system related complications at the end of the procedure.
Time Frame: Within 30 days of implant procedure
Population: Analysis for this endpoint includes subjects with an implant attempt.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Engager™ Aortic Valve
Number analyzed (Participants) | 20
percentage of participants | 95.0 [75.1 to 99.9]

2. Other Pre Specified Outcome: Device Success According to VARC2
Description: Device success is a composite of:
  Absence of 30-day in-hospital death Correct position of the device within the aortic annular region Intended performance of the bioprosthesis (no patient-prosthesis mismatch, mean aortic gradient <20 mmHg or peak velocity <3 m/s at discharge, and no moderate or severe prosthetic valve regurgitation)
Time Frame: 30 days post-procedure
Population: Analysis for this endpoint includes subjects with an implant attempt.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Engager™ Aortic Valve
Number analyzed (Participants) | 20.0
percentage of participants | 15.0 [3.2 to 37.9]

3. Other Pre Specified Outcome: Composite 30-day Safety Endpoint According to VARC2
Description: Percentage of Participants with any of the following Safety Events within 30-days post-procedure:
  All-cause mortality All stroke Life-threatening bleeding Acute kidney injury (stage 2-3) Coronary artery obstruction requiring intervention Major vascular complication Valve-related dysfunction requiring repeat procedure (BAV, TAVI or SAVR)
Time Frame: 30-days post-procedure
Population: Analysis for this endpoint includes subjects with an implant attempt.
Measure: Number; unit: percentage of participants
Arm/Group | Engager™ Aortic Valve
Number analyzed (Participants) | 20
percentage of participants | 25.0

4. Other Pre Specified Outcome: Composite Clinical Efficacy Endpoint After 30 Days According to VARC2
Description: Percentage of Participants with any of the following Safety Events after 30-days post-procedure:
  All-cause mortality All stroke Hospitalization for valve-related symptoms or worsening congestive heart failure
Time Frame: 30-days post-procedure
Population: Analysis for this endpoint includes subjects at risk (or alive and in study) at 30 days.
Measure: Number; unit: percentage of participants
Arm/Group | Engager™ Aortic Valve
Number analyzed (Participants) | 18
percentage of participants | 94.4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 1 year post-implant procedure.
Description: SAEs were adjudicated per VARC2 definitions.
Arm/Group | Engager™ Aortic Valve
Serious Adverse Events (participants affected / at risk) | 20/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engager™ Aortic Valve (N=20)
Anemia (Hgb<10g or Hct<30%) (Blood and lymphatic system disorders) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Congestive heart failure (Cardiac disorders) | 3 (3)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrio-ventricular block, 3 degree (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Other implantation/catheterization (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Other cardiac event (Cardiac disorders) | 1 (1)
Life threatening or disabling bleed event (Gastrointestinal disorders) | 1 (1)
Major bleeding event (Gastrointestinal disorders) | 1 (1)
Other gastrointestinal (Gastrointestinal disorders) | 2 (2)
Multi organ failure (General disorders) | 1 (1)
Other (General disorders) | 1 (1)
Sepsis, confirmed (positive blood culture) (General disorders) | 1 (1)
Other gastrointestinal (Infections and infestations) | 1 (1)
Life threatening or disabling bleed event (Injury, poisoning and procedural complications) | 1 (1)
Major bleeding event (Injury, poisoning and procedural complications) | 1 (1)
Misplacement of the Engager Valve (Injury, poisoning and procedural complications) | 1 (1)
Other (Injury, poisoning and procedural complications) | 1 (1)
Perforation of the heart (Injury, poisoning and procedural complications) | 2 (2)
Other (Investigations) | 1 (1)
Cancer/malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Other (Psychiatric disorders) | 1 (1)
Acute kidney injury: stage 3 (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Life threatening or disabling bleed event (Surgical and medical procedures) | 1 (1)
Major ascending aortic dissection (Vascular disorders) | 1 (1)
Other (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engager™ Aortic Valve (N=20)
Anemia (Hgb<10g or Hct<30%) (Blood and lymphatic system disorders) | 3 (3)
Hemolysis: minor (Blood and lymphatic system disorders) | 1 (1)
Other hematologic/oncologic (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrio-ventricular block, 1 degree (Cardiac disorders) | 2 (2)
Congestive heart failure (Cardiac disorders) | 1 (1)
LBBB (Cardiac disorders) | 3 (3)
Other arrhythmia (Cardiac disorders) | 1 (1)
Other respiratory/pulmonary (Cardiac disorders) | 1 (1)
Pericardial effusion, non-hemorrhagic (Cardiac disorders) | 1 (1)
Sinus bradycardia (<50 bpm) (Cardiac disorders) | 2 (2)
Ventricular premature beats (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Other (Endocrine disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Minor bleeding event (Gastrointestinal disorders) | 1 (1)
Other (Gastrointestinal disorders) | 2 (4)
Other gastrointestinal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Other (General disorders) | 3 (3)
Other (Infections and infestations) | 1 (1)
Other infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3)
Other (Injury, poisoning and procedural complications) | 2 (3)
Congestive heart failure (Investigations) | 1 (1)
Other (Investigations) | 3 (3)
Other gastrointestinal (Investigations) | 1 (1)
Other renal (Investigations) | 1 (1)
Other (Metabolism and nutrition disorders) | 1 (2)
Other (Musculoskeletal and connective tissue disorders) | 4 (4)
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Other central nervous system (Nervous system disorders) | 1 (1)
Other (Psychiatric disorders) | 4 (4)
Other (Renal and urinary disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm/asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Minor bleeding event (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Other respiratory/pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other (Skin and subcutaneous tissue disorders) | 3 (3)
Other (Vascular disorders) | 2 (2)
Other cardiac event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less